CLINICAL TRIAL: NCT01680198
Title: Effect of Paricalcitol on Endothelial Function in Chronic Kidney Disease (CKD) Patients (the PENNY Study)
Brief Title: Paricalcitol and Endothelial Function in Chronic Kidney Disease Patients (the PENNY Study)
Acronym: PENNY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Carmine Zoccali, Prof., Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oct2010PENNYStudy
Record Dates: First submitted 2012-08-30; First posted 2012-09-07 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Kidney Disease.
Keywords: Vitamin D; Paracalcitol; Chronic kidney disease; Endothelial dysfunction; Flow mediated vasodilation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules daily for 12 weeks.
  Interventions: Drug: placebo
- Paracalcitol (Experimental): see "Intervention description" for details.
  Interventions: Drug: Paracalcitol

INTERVENTIONS:
Drug: Paracalcitol — Patients in the experimental arm received 2 micrograms Paricalcitol capsules daily, for 12 weeks. This dose was adjusted based on clinical laboratory parameters and the maximum dose was 2 micrograms daily.
  Other Names: Active form of Vitamin D.
  Arms: Paracalcitol
Drug: placebo
  Arms: Placebo

SUMMARY:
The primary aim of this study was to test the hypothesis that Paricalcitol, an active form of vitamin D, improved endothelial function in stage 3-4 chronic kidney disease (CKD) patients. A secondary aim of this trial was to study the relationship between endothelial function and plasma/serum and genetic biomarkers of bone mineral disorders in CKD (BMD-CKD) and renin angiotensin-aldosteron system (RAS) (angiotensin II and plasma renin activity).

DETAILED DESCRIPTION:
Primary objective: Test the hypothesis that Paricalcitol, an active form of vitamin D improves endothelial function in stage 3-4 chronic kidney disease (CKD) patients.

Secondary analysis: Study the relationship between endothelial function and plasma/serum and genetic biomarkers of bone mineral disorders in CKD (BMD-CKD) and renin angiotensin-aldosteron system (RAS) (angiotensin II and plasma renin activity).

Background:

Endothelial function is altered in patients with CKD. Factors responsible for disturbed endothelium-dependent vasodilatation in CKD include reduced bioactivity of the nitric oxide (NO) pathway with decreased endothelial NO synthase (NOS) activity or inhibition via accumulation of endogenous inhibitors. In patients with CKD and in those on dialysis serum 25(OH)D3 and 1,25(OH)2D3 levels are associated with FMD. Vitamin D receptors and 1 -hydroxylase activity are present in endothelial and vascular smooth muscle cells and 1,25(OH)2D3 stimulates vascular endothelial growth factor and prostacyclin production by vascular smooth muscle cells. These biological observations may have clinical implications because paricalcitol treatment predicts longer survival in ESRD patients and very recent data link vitamin D to progression to ESRD in patients with stage 3-5 CKD. Furthermore, a previous study by us has shown that the BMSI polymorphism of the vitamin D receptor gene is associated with LVH and LVH progression in ESRD patients.

Study population: Patients with stage 3-4 CKD of both sexes in the age range 18-80 years. Patients taking vitamin D supplements, with abnormal liver function tests, symptomatic cardiovascular disease, diabetes or cancer and those whose medications changed during the study were excluded.

Design and Methods: The study was a double-blind, randomized, parallel groups trial. After baseline measurements, patients with iPTH level > 65 pg/ml; Ca between 8.4- 10.00 mg/dL and P between 2.9-4.5 were randomized to receive 2 micrograms Paricalcitol capsules (or matching placebo) daily, for 12 weeks. This doses was adjusted based on clinical laboratory parameters and the maximum dose was 2 micrograms daily.

During the study if a subject experienced over suppression of serum iPTH (defined as a serum iPTH <15 pg/mL), or hypercalcemia (defined as Ca > 11.0 mg/dL), the subject continued to take study drug at reduced dosage 1 mcg any other day and returned in 2 weeks for an unscheduled visit. If the values from the unscheduled visit serum iPTH and/or Ca did not returned to > 15 pg/mL and/or <11.0 mg/dL, respectively, the drug was discontinued.

Flow mediated vasodilatation was measured according to a validated protocol developed at the coordinating center of a national (Italian)working group of vascular function testing.

Primary end-point: Change in Flow Mediated Dilatation (FMD) induced by Paricalcitol in comparison to Placebo.

Study power: To detect a 2% difference (standard deviation: ± 3.0%) in the change in FMD between Paracalcitol treated and untreated patients with a power of 80 %, a confidence level using a two-tailed test of 5% and a potential attrition rate of 15%, at least 44 patients per group were required (88 patients in total).

Statistical analysis: Data will be summarized as mean ± standard deviation (normally distributed data), median and inter-quartile range (non normally distributed data) or as percent frequency, and comparison between groups will be made by independent T-Test, Mann-Whitney Test, or Chi Square test, as appropriate. Within patients comparisons will be done by statistical tests for paired observations. Data analysis of the primary outcome will be performed by comparing the changes in FMD in Paracalcitol treated and untreated patients by using the T-Test for independent observations. Possible differences in risk factors at baseline not controlled by randomization (i.e. differences due to chance) will be accounted for by using multivariate regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with iPTH level > 65 pg/ml; Ca between 8.4- 10.00 mg/dL and P between 2.9-4.5
* Negative serum pregnancy test for female subjects of childbering potential.
* Informed consent.

Exclusion Criteria:

* Use vitamin D supplements.
* Altered liver function tests (bilirubin, aminotransferases and total alkaline phosphatase > 3 times the upper limit of normal ranges).
* Sympthomatic cardiovascular disease on the basis of clinical history. Cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Endothelial function measurement | 12 weeks from baseline
  Endothelial-dependent and independent vasodilation was assessed by a Toshiba Nemia XG Echo-Doppler applying a 7.5 MHz transducer that was fixed by an adjustable stereotactic clamp to warrant image stability. After baseline recording (1 min) a standard sphygmomanometer was placed on the right forearm 2 cm below the elbow and the cuff was inflated to 250 mmHg for 5 min. Recordings were performed during the 4 min following cuff deflation to estimate endothelium-dependent FMD. In studies of endothelium-independent vasodilatation recording times were 1 min for the baseline assessment and 5 min for changes in arterial diameter brought about by GTN. An interval of at least 1h was set between the last FMD assessment and GTN administration. All scans were recorded, stored and analyzed off-line. FMD and GTN were computed as the maximal % increase in diameter over baseline by an automatic edge detection system.

SECONDARY OUTCOMES:
Endothelial function and plasma/serum and genetic biomarkers of bone mineral disorders in CKD (BMD-CKD) and renin angiotensin-aldosteron system (RAS). | 12 weeks from baseline
  The investigators will analyze the relationship between endothelial function and plasma/serum and genetic biomarkers of bone mineral disorders in CKD (BMD-CKD) and renin angiotensin-aldosteron system (RAS) (angiotensin II and plasma renin activity).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Curatola, MD, Study Director — Nephrology, Dialysis and Transplantation Unit
Locations (1):
- Nephrology, Dialysis and Transplantation Unit, Reggio Calabria, Reggio Calabria, Italy

REFERENCES:
- [Background] Yilmaz MI, Sonmez A, Saglam M, Yaman H, Kilic S, Demirkaya E, Eyileten T, Caglar K, Oguz Y, Vural A, Yenicesu M, Zoccali C. FGF-23 and vascular dysfunction in patients with stage 3 and 4 chronic kidney disease. Kidney Int. 2010 Oct;78(7):679-85. doi: 10.1038/ki.2010.194. Epub 2010 Jul 7. PMID 20613714
- [Background] London GM, Guerin AP, Verbeke FH, Pannier B, Boutouyrie P, Marchais SJ, Metivier F. Mineral metabolism and arterial functions in end-stage renal disease: potential role of 25-hydroxyvitamin D deficiency. J Am Soc Nephrol. 2007 Feb;18(2):613-20. doi: 10.1681/ASN.2006060573. Epub 2007 Jan 3. PMID 17202417
- [Background] Yamamoto T, Kozawa O, Tanabe K, Akamatsu S, Matsuno H, Dohi S, Hirose H, Uematsu T. 1,25-dihydroxyvitamin D3 stimulates vascular endothelial growth factor release in aortic smooth muscle cells: role of p38 mitogen-activated protein kinase. Arch Biochem Biophys. 2002 Feb 1;398(1):1-6. doi: 10.1006/abbi.2001.2632. PMID 11811942
- [Background] Wakasugi M, Noguchi T, Inoue M, Kazama Y, Tawata M, Kanemaru Y, Onaya T. Vitamin D3 stimulates the production of prostacyclin by vascular smooth muscle cells. Prostaglandins. 1991 Aug;42(2):127-36. doi: 10.1016/0090-6980(91)90072-n. PMID 1775635
- [Background] Teng M, Wolf M, Ofsthun MN, Lazarus JM, Hernan MA, Camargo CA Jr, Thadhani R. Activated injectable vitamin D and hemodialysis survival: a historical cohort study. J Am Soc Nephrol. 2005 Apr;16(4):1115-25. doi: 10.1681/ASN.2004070573. Epub 2005 Feb 23. PMID 15728786
- [Background] Teng M, Wolf M, Lowrie E, Ofsthun N, Lazarus JM, Thadhani R. Survival of patients undergoing hemodialysis with paricalcitol or calcitriol therapy. N Engl J Med. 2003 Jul 31;349(5):446-56. doi: 10.1056/NEJMoa022536. PMID 12890843
- [Background] Ravani P, Malberti F, Tripepi G, Pecchini P, Cutrupi S, Pizzini P, Mallamaci F, Zoccali C. Vitamin D levels and patient outcome in chronic kidney disease. Kidney Int. 2009 Jan;75(1):88-95. doi: 10.1038/ki.2008.501. Epub 2008 Oct 8. PMID 18843258
- [Background] Testa A, Mallamaci F, Benedetto FA, Pisano A, Tripepi G, Malatino L, Thadhani R, Zoccali C. Vitamin D receptor (VDR) gene polymorphism is associated with left ventricular (LV) mass and predicts left ventricular hypertrophy (LVH) progression in end-stage renal disease (ESRD) patients. J Bone Miner Res. 2010 Feb;25(2):313-9. doi: 10.1359/jbmr.090717. PMID 20422622
- [Background] Ghiadoni L, Faita F, Salvetti M, Cordiano C, Biggi A, Puato M, Di Monaco A, De Siati L, Volpe M, Ambrosio G, Gemignani V, Muiesan ML, Taddei S, Lanza GA, Cosentino F. Assessment of flow-mediated dilation reproducibility: a nationwide multicenter study. J Hypertens. 2012 Jul;30(7):1399-405. doi: 10.1097/HJH.0b013e328353f222. PMID 22525207
- [Derived] D'arrigo G, Pizzini P, Cutrupi S, Tripepi R, Tripepi G, Mallamaci F, Zoccali C. Vitamin D receptor activation raises soluble thrombomodulin levels in chronic kidney disease patients: a double blind, randomized trial. Nephrol Dial Transplant. 2019 May 1;34(5):819-824. doi: 10.1093/ndt/gfy085. PMID 29668990
- [Derived] Torino C, Pizzini P, Cutrupi S, Tripepi R, Vilasi A, Tripepi G, Mallamaci F, Zoccali C. Effect of Vitamin D Receptor Activation on the AGE/RAGE System and Myeloperoxidase in Chronic Kidney Disease Patients. Oxid Med Cell Longev. 2017;2017:2801324. doi: 10.1155/2017/2801324. Epub 2017 Dec 6. PMID 29362665
- [Derived] Spoto B, Pizzini P, Tripepi G, Mallamaci F, Zoccali C. Circulating adiponectin modifies the FGF23 response to vitamin D receptor activation: a post hoc analysis of a double-blind, randomized clinical trial. Nephrol Dial Transplant. 2018 Oct 1;33(10):1764-1769. doi: 10.1093/ndt/gfx344. PMID 29304245
- [Derived] Zoccali C, Curatola G, Panuccio V, Tripepi R, Pizzini P, Versace M, Bolignano D, Cutrupi S, Politi R, Tripepi G, Ghiadoni L, Thadhani R, Mallamaci F. Paricalcitol and endothelial function in chronic kidney disease trial. Hypertension. 2014 Nov;64(5):1005-11. doi: 10.1161/HYPERTENSIONAHA.114.03748. Epub 2014 Aug 4. PMID 25259743